CLINICAL TRIAL: NCT04272125
Title: Safety and Efficacy of CD123-Targeted CAR-T Therapy for Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC016
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute
Keywords: Leukemia; Acute Myeloid Leukemia; CD123; CAR-T
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD123 CAR-T cells treat (Experimental): Patients will be be treated with CD123 CAR-T cells
  Interventions: Biological: CD123 CAR-T cells

INTERVENTIONS:
Biological: CD123 CAR-T cells — A single infusion of CD123-CAR-T cells will be administered intravenously

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of CD123-targeted CAR-T cells therapy for patients with relapsed/refractory Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
There are limited options for treatment of relapse/refractory Acute Myeloid Leukemia. CD123 is expressed on most myeloid leukemia cells so it is an ideal target for CAR-T. Some researches have revealed that CD123 is a marker of leukemia stem cells, which indicates that the eradication of CD123 cells may prevent relapse of leukemia. In this study, investigators will evaluate the safety and efficacy of CAR-T targeting CD123 in patients with relapsed/refractory Acute Myeloid Leukemia. The primary goal is safety and efficiency assessment, including adverse events and disease status after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Diagnose as relapsed /refractory acute myeloid leukemia, and meet one of the following conditions:

   1. Failed to standard chemotherapy regimens;
   2. Relapse after complete remission, high-risk and / or refractory patients ;
   3. Relapse after hematopoietic stem cell transplantation;
3. Evidence for cell membrane CD123 expression;
4. All genders, ages: 3 to 75 years；
5. The expect time of survive is above 12 weeks;
6. KPS>60；
7. No serious mental disorders ;
8. Left ventricular ejection fraction ≥50%
9. Sufficient hepatic function defined by ALT/AST≤3 x ULN and bilirubin≤2 x ULN;
10. Sufficient renal function defined by creatinine clearance≤2 x ULN;
11. Sufficient pulmonary function defined by indoor oxygen saturation≥92%;
12. With single or venous blood collection standards, and no other cell collection contraindications;
13. Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Have received CAR-T therapy or other genetically modified cell therapy before screening；
2. Participated in other clinical research within 1 month before screening；
3. Have received the following anti-tumor treatment before screening: Have received chemotherapy, targeted therapy or other experimental drug treatment within 4 weeks, except those who have confirmed disease progression after treatment;
4. Live attenuated vaccine within 4 weeks before screening;
5. Convulsion or stoke within past 6 months;
6. Previous history of other malignancy;
7. Presence of uncontrolled active infection;
8. Subjects with positive HBsAg or HBcAb positive and peripheral blood HBV DNA titer is higher than the lower limit of detection of the research institution; HCV antibody positive and peripheral blood HCV RNA titer is higher than the lower limit of detection of the research institution; HIV antibody positive; syphilis primary screening antibody positive;
9. Pregnant or breasting-feeding women;
10. Any situation that investigators regard not suitable for attending in this study or may affect the data analysis.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The response rate of CD123 CAR-T treatment in patients with relapse/refractory Acute Myeloid Leukemia that treatment by CD123 CAR-T cells therapy | 6 months
  The response rate of CD123 CAR-T treatment will be recorded and assessed according to the National Comprehensive Cancer Network Guideline

SECONDARY OUTCOMES:
Rate of CD123 CAR-T cells in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) rate of CD123 CAR-T cells were determined by means of flow cytometry
Quantity of CD123 CAR copies in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) quantity of CD123 CAR copies were determined by means of qPCR
Cellular kinetics of CD123 positive cells in bone marrow | 1 years
  In vivo (bone marrow) rate and quantity of CD123 positive cells were determined by means of flow cytometry
Levels of cytokines in serum | 3 months
  In vivo (serum) quantity of cytokines
Duration of Response (DOR) of CD123 CAR-T treatment in patients with refractory/relapsed acute myeloid leukemia | 2 years
  DOR will be assessed from the first assessment of CR/CRi to the first assessment of recurrence or progression of the disease or death from any cause (censored)
Progress-free survival(PFS) of CD123 CAR-T treatment in patients with refractory/relapsed acute myeloid leukemia | 2 year
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression (censored)
Overall survival(OS) of CD123 CAR-T treatment in patients with refractory/relapsed acute myeloid leukemia | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause (censored)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Qian, PhD, Principal Investigator — Chongqing University Cancer Hospital; Ying Xiang, MD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China